CLINICAL TRIAL: NCT01255891
Title: A Phase II Study of Adjuvant Androgen Suppression Plus Radiation Therapy for High-Risk Localized Adenocarcinoma of the Prostate
Brief Title: Adjuvant Androgen Suppression Plus Radiation Therapy for High-Risk Localized Adenocarcinoma Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Tamim Niazi (Other)
Collaborators: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor-Investigator, Dr. Tamim Niazi, Principal Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Organization: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: McG 0913
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: high risk localized adenocarcinoma of the prostate
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- Adjuvant (Other): Adjuvant suppression plus radiation therapy
  Interventions: Radiation: Androgen suppression plus radiation therapy

INTERVENTIONS:
Radiation: Androgen suppression plus radiation therapy — Adjuvant androgen suppression plus radiation therapy

SUMMARY:
To evaluate the efficacy of LHRH agonist with adjuvant pelvic radiation therapy in post radical prostatectomy patients with high risk pathological features for failure. To determine the freedom from biochemical (maintenance of a PSA less than nadir + 2 ng/ml) and clinical progression rate at 5 years.

DETAILED DESCRIPTION:
Same as brief Summary

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma of the prostate treated primarily with radical prostatectomy, pathologically proven to be lymph node negative by pelvic lymphadenectomy (N0) or lymph node status pathologically unknown (undissected pelvic lymph nodes [Nx]), i.e. lymph node dissection is not required;
2. Any type of radical prostatectomy will be permitted, including retropubic, perineal laparoscopic or robotically assisted. If performed, the number of lymph nodes removed per side of the pelvis and the extent of the pelvic lymph node dissection (obturator vs. extended lymph node dissection) should be noted. There is no time limit for the date of radical prostatectomy.
3. A post-radical prostatectomy entry PSA of > 0 and < 1 ng/ml at least 6 weeks after prostatectomy and within 30 days of registration.
4. One of the following pathologic/chemical classifications:

   * T3N0/Nx disease with or without positive surgical margin; or;
   * Gleason score of 8 or more;
   * Pre prostatectomy PSA > 20 ng/ml
5. KPS > 70
6. Age ≥ 18;
7. No distant metastases, based upon the following minimum diagnostic workup:
8. History/physical examination (including digital rectal exam) within 8 wks prior to registration;
9. A CT scan or MRI of the abdomen and pelvis within 120 days prior to registration;
10. Bone scan within 120 days prior to registration; if the bone scan is suspicious, a plain x-ray and/or MRI must be obtained to rule out metastasis.
11. Adequate bone marrow function, within 90 days prior to registration, defined as follows:

    * Platelets ≥ 100,000 cells/mm3 based upon CBC;
    * Hemoglobin ≥ 10.0 g/dl based upon CBC
    * AST or ALT < 2 x the upper limit of normal within 90 days prior to registration;
12. Patients must sign a study-specific informed consent prior to study entry.

EXCLUSION CRITERIA:

1. A palpable prostatic fossa abnormality/mass suggestive of recurrence, unless shown by biopsy under ultrasound guidance not to contain cancer;
2. N1 patients are ineligible, as are those with pelvic lymph node enlargement ≥ 1.5 cm in greatest dimension by CT scan or MRI of the pelvis, unless the enlarged lymph node is sampled and is negative;
3. Androgen deprivation therapy started prior to prostatectomy for > 6 months duration;
4. Androgen deprivation therapy started after prostatectomy and prior to registration;
5. Prior pelvic radiotherapy;
6. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 5 years (for example, carcinoma in situ of the oral cavity is permissible);
7. Severe, active co-morbidity, defined as follows:

   * History of inflammatory bowel disease;
   * History of hepatitis B or C; Blood tests are not required to determine if the patient has had hepatitis B or C, unless the patient reports a history of hepatitis.
   * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
   * Transmural myocardial infarction within the last 6 months
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
   * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration;
   * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; AST or ALT are required; note, however, that laboratory tests for coagulation parameters are not required for entry into this protocol.
   * Prior allergic reaction to the study drug(s) involved in this protocol.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-01; Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
to determine the rate of local and distance failure at 5 years | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tamim Niazi, MD, Principal Investigator — McGill University Department of Oncology
Locations (2):
- Canada (2):
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Elakshar S, Tolba M, Tisseverasinghe S, Pruneau L, Di Lalla V, Bahoric B, Niazi T. Salvage Whole-Pelvic Radiation and Long-Term Androgen-Deprivation Therapy in the Management of High-Risk Prostate Cancer: Long-Term Update of the McGill 0913 Study. Curr Oncol. 2023 Aug 1;30(8):7252-7262. doi: 10.3390/curroncol30080526. PMID 37623007
- [Derived] Kucharczyk MJ, Tsui JMG, Khosrow-Khavar F, Bahoric B, Souhami L, Anidjar M, Probst S, Chaddad A, Sargos P, Niazi T. Combined Long-Term Androgen Deprivation and Pelvic Radiotherapy in the Post-operative Management of Pathologically Defined High-Risk Prostate Cancer Patients: Results of the Prospective Phase II McGill 0913 Study. Front Oncol. 2020 Mar 12;10:312. doi: 10.3389/fonc.2020.00312. eCollection 2020. PMID 32226774